CLINICAL TRIAL: NCT05222360
Title: Improvement of Body Image Flexibility in High School Female Athletes Undergoing Three Educational Sessions About Nutrition and Body Image
Brief Title: Improvement of Body Image Flexibility in High School Female Athletes Doing Educational About Nutrition and Body Image
Status: Completed | Type: Observational
Sponsor: Rocky Mountain Sports Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 52345
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Body Image; Nutrition, Healthy
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female high school athletes: Athletes who identify as female at a local high school who are in an athletic program. There was no control group as the school wanted everyone to have the 3 educational sessions. The athletes underwent 3 educational sessions. No medication was used. Education was the intervention
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — 3 educational sessions about body image and nutrition

SUMMARY:
Evaluation of increase in body flexibility in female high school athletes undergoing education on nutrition and body image

DETAILED DESCRIPTION:
This study was a prospective cohort design. Female high school athletes were asked to participate in three educational sessions about nutrition, body image flexibility, and RED-S (relative energy deficiency in sport). Pre and post-tests were done with a validated tool measuring body image flexibility.

ELIGIBILITY:
Inclusion Criteria:

* identify as female
* athlete at local high school
* willing to fill out survey at beginning and end of sessions
* willing to provide consent

Exclusion Criteria:

* none

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — identify as female
Study Population: These are athletes at local high schools who identify as female. The demographic area is primarily socioeconomically middle class.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
BI-AAQ Scores | 2 months
  scores on body image flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Vidlock, M.D., Principal Investigator — Rocky Mountain Sports Medicine
Locations (1):
- Rocky Mountain Sports Medicine, Parker, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
We have yet to find a place that shares BI-AAQ data as it is a unique questionaire